CLINICAL TRIAL: NCT06605534
Title: LEAD Pilot Study: Leveraging the Emergency Department to Address SDOH and Reduce Lung Cancer Screening Disparities
Brief Title: Leveraging the Emergency Department (LEAD) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: New Jersey Commission on Cancer Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Pro2024-0236
Record Dates: First submitted 2024-09-11; First posted 2024-09-20 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Lung Cancer
Keywords: screening; lung cancer; Disparities; social determinants of health; emergency department
MeSH Terms: conditions — Lung Neoplasms; Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LungTalk Group (Experimental): LungTalk is a novel theoretically grounded health educational tool that will be delivered via iPad and is an interactive computer-based program that includes audio, video and animation segments with scripts presented from a master content library in consideration of different ways people like to learn. Informed by our prior research, LungTalk tailors its content based on smoking status and perceived barriers. In prior work, LungTalk more than doubled Lung Cancer Screening (LCS) knowledge and health beliefs (p < 0.01), and was associated with a significant increase in deciding to screen for lung cancer compared to control group; OR 1.99; 95% CI, 1.03, 3.85, p = 0.03.
  Interventions: Behavioral: LungTalk
- Non-tailored Lung Screening Pamphlet Group (Active Comparator): Non-tailored Lung Screening Pamphlet is a non-tailored educational brochure, What is Lung Cancer Screening from the GO2 Foundation that will be emailed to the patient. This widely used educational standard of care is a 2-page reader-friendly non-tailored electronic brochure about risk and screening for lung cancer used in clinical and community settings.
  Interventions: Other: Non-tailored lung screening

INTERVENTIONS:
Behavioral: LungTalk — Tailored lung screening intervention
  Arms: LungTalk Group
Other: Non-tailored lung screening — Non-tailored lung screening. It involves the addition of education to Social Determinants of Health (SDOH) screening and referral with patient navigation. Patients will be identified, and screened for SDOH needs using the UniteUs SDOH screener that is embedded in the Electronic Health Record (EHR), and connected to geographically-tailored resources (as described above under Arm 1). Participants will then be sent a non-tailored lung screening educational brochure via email to review that details lung cancer risk, lung screening facts, benefits, and potential harms. Within 48 hours, the Community Outreach and Engagement (COE) Patient Navigator will contact the patient to answer questions and provide navigation services as described above in Arm 1.
  Arms: Non-tailored Lung Screening Pamphlet Group

SUMMARY:
This is a pilot Type 1 Hybrid Effectiveness-Implementation Trial. The study will first examine reach in a non-traditional setting (the Emergency Department - ED) that uses an Electronic Health Record (EHR)-embedded Social Determinants of Health (SDoH) screening tool to identify lung screening-eligible patients for a tailored intervention to increase lung screening uptake. Reach is defined as the absolute number, proportion, and representativeness of individuals targeted for lung screening knowledge, awareness, and uptake. Then, a pilot trial will be conducted to examine the preliminary effectiveness of a tailored lung screening intervention compared to enhanced usual care to influence individual-level potential drivers of lung screening (health literacy, mistrust, stigma, fatalism, knowledge, lung screening health beliefs) and the ability to increase lung screening uptake among screening-eligible patients. Quantitative (Randomized Controlled Trial and EHR data) methods will be used for data collection and analysis to address the study aims.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years to 80 years
* Currently smoke cigarettes or quit smoking cigarettes within the past 15 years
* 20 pack-year smoking history
* Has never had lung cancer screening
* Able to provide informed consent
* Able to speak and understand English

Exclusion Criteria:

* Diagnosed with lung cancer
* Has a history of having a lung cancer screening scan
* Unable to speak and understand English

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Lung Cancer Screening Uptake | Assessed at 1 month and 6 months post intervention
  Completion of a Screening Low-Dose Computed Tomography (LDCT) of the Chest confirmed via Electronic Health Records (EHR))
Stage of Adoption for Lung Cancer Screening | Assessed at 1 week and then at 1 month and 6 months post intervention
  Screening Intention will be assessed with the Stage of Adoption for Decision- Making About Lung Screening using an algorithm of questions used in our prior studies assessing the 7 stages (unaware, aware but unengaged, undecided, decided not to act, decided to act, action, and maintenance). This will allow investigators to assess intent.

SECONDARY OUTCOMES:
Health Literacy Scale | At one week and one month post intervention
  Change in Health Literacy Scale between baseline and 1 week and 1-month post-intervention. The Health Literacy Scale will be measured using the 3-item psychometrically validated Health Literacy Scale by Chew and colleagues. This scale has been supported as valid for detecting inadequate health literacy using Likert scale response options ranging from 0=strongly disagree to 4 =strongly agree with lower scores representative of higher levels of health literacy.
Medical Mistrust Scale | At one week and one month post intervention
  Change in Medical Mistrust Scale between baseline and 1 week and 1-month post-intervention. Medical Mistrust will be measured using the psychometrically validated 5-item Medical Mistrust Scale. This measure assesses constructs related to mistrust of the medical system, including suspicion, discrimination, and lack of support. Likert scale response options range from 1 to 4 with 1=Stongly Disagree to Agree 5=Strongly. Responses are summed (range 5-25), with higher scores indicating more trust. *Negatively worded item is reverse coded. Reliability and validity have been well established with Cronbach's alpha of 0.87-0.88.
Perceived Stigma Scale | At one week and one month post intervention
  Change in Perceived Stigma Scale between baseline and 1 week and 1-month post-intervention. Perceived Stigma will be measured using the 5-item smoking-related stigma subscale of the Cataldo Lung Cancer Stigma Scale. The response scale is 1=strongly disagree to 4=strongly agree; range is 5 to 25 (higher stigma). Cronbach's alphas were 0.75 to 0.89 in prior studies.
Perceived Risk of Lung Cancer Scale | At one week and one month post intervention
  Change in Perceived Risk of Lung Cancer Scale between baseline and 1 week and 1-month post-intervention. Lung Cancer Screening Health Belief Scales will be used to measure perceived risk, perceived benefits, perceived barriers, and self-efficacy. Content and construct validity have been established. Internal consistency reliability was established by our team with a sample of 497 lung cancer screening-eligible individuals with Perceived Risk of Lung Cancer on a 3-item scale with Likert-type responses from 1=Strongly Disagree to 4=Strongly Agree. The range of scores is 3 to 12 (higher perceived risk of lung cancer). Cronbach's alpha was 0.88 in our preliminary study.
Perceived Benefits of Lung Cancer Screening Scale | At one week and one month post intervention
  Change in Perceived Benefits of Lung Cancer Screening Scale between baseline and 1 week and 1-month post-intervention. Lung Cancer Screening Health Belief Scales will be used to measure perceived risk, perceived benefits, perceived barriers, and self-efficacy. Content and construct validity have been established. Internal consistency reliability was established by our team with a sample of 497 lung cancer screening-eligible individuals with Perceived Benefits of Lung Cancer Screening on a 6-item scale with responses ranging from 1=strongly disagree to 4=strongly agree. The range of scores is 6 to 24 (higher perceived benefits), with a Cronbach's alpha of 0.76 in our preliminary study
Perceived Barriers to Lung Cancer Screening Scale | At one week and one month post intervention
  Change in Perceived Barriers of Lung Cancer Screening Scale between baseline and 1 week and 1-month post-intervention. Lung Cancer Screening Health Belief Scales will be used to measure perceived risk, perceived benefits, perceived barriers, and self-efficacy. Content and construct validity have been established. Internal consistency reliability was established by our team with a sample of 497 lung cancer screening-eligible individuals with Perceived Barriers to Lung Cancer Screening. This scale has 17 items with four-point Likert responses where 1=strongly disagree and 4=strongly agree. The range of scores is 17 to 68 (higher perceived barriers) with a Cronbach's a of 0.87 in our preliminary psychometric study
Self-Efficacy for Lung Cancer Screening Scale | At one week and one month post intervention
  Change in Self-Efficacy for Lung Cancer Screening Scale between baseline and 1 week and 1-month post-intervention. Lung Cancer Screening Health Belief Scales will be used to measure perceived risk, perceived benefits, perceived barriers, and self-efficacy. Content and construct validity have been established. Internal consistency reliability was established by our team with a sample of 497 lung cancer screening-eligible individuals with Self-Efficacy for Lung Cancer Screening. This scale has nine items with a four-point Likert response option (1=Not at all Confident and 4 =Very Confident) to assess individual beliefs about ability to arrange and complete an LDCT to screen for lung cancer. The range of scores is 9 to 36 (higher levels of self-efficacy) with a Cronbach's alpha of 0.92 in our preliminary psychometric study.
Knowledge: Lung Cancer and Screening Scale | At one week and one month post intervention
  Change in Knowledge: Lung Cancer and Lung Screening between baseline and 1 week and 1-month post-intervention. Knowledge of Lung Cancer and Lung Screening will be assessed with a 7-item multidimensional scale used in our preliminary studies adapted from literature specific to lung cancer. Several aspects will be assessed, including knowledge of lung cancer, risk, and screening. The range of scores is 0 to 7, with 0 being No Knowledge, and 9 being Complete Knowledge.
Lung Cancer Fatalism | At one week and one month post intervention
  Change in Lung Cancer Fatalism between baseline and 1 week and 1-month post-intervention. Lung Cancer Fatalism will be measured with the 11-item dichotomous (0=yes and 1=no) Lung Cancer Fatalism Scale adapted from the Revised Powe Fatalism Inventory that has been psychometrically validated.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Carter-Bawa, PhD, Principal Investigator — Hackensack Meridian Health
Locations (10):
- United States (10):
  - Ocean Medical Center, Brick, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Bayshore Medical Center, Holmdel, New Jersey
  - Southern Ocean Medical Center, Manahawkin, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Palisades Medical Center, North Bergen, New Jersey
  - Old Bridge Medical Center, Old Bridge, New Jersey
  - Raritan Bay Medical Center, Perth Amboy, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] Cancer Facts & Figures for African Americans 2019-2021. In: American Cancer Society. Atlanta: 2019.
- [Background] United States Preventive Services Task Force. Final recommendation statement: Lung cancer screening.http://www.uspreventiveservicestaskforce.org/Page/Document/RecommendationStatem entFinal/lung-cancer-screening. Updated December 2016. Accessed January 21, 2023.
- [Background] Rivera MP, Katki HA, Tanner NT, Triplette M, Sakoda LC, Wiener RS, Cardarelli R, Carter-Harris L, Crothers K, Fathi JT, Ford ME, Smith R, Winn RA, Wisnivesky JP, Henderson LM, Aldrich MC. Addressing Disparities in Lung Cancer Screening Eligibility and Healthcare Access. An Official American Thoracic Society Statement. Am J Respir Crit Care Med. 2020 Oct 1;202(7):e95-e112. doi: 10.1164/rccm.202008-3053ST. PMID 33000953
- [Background] Carter-Harris L, Tan AS, Salloum RG, Young-Wolff KC. Patient-provider discussions about lung cancer screening pre- and post-guidelines: Health Information National Trends Survey (HINTS). Patient Educ Couns. 2016 Nov;99(11):1772-1777. doi: 10.1016/j.pec.2016.05.014. Epub 2016 May 17. PMID 27241830
- [Background] American Lung Association: State of Lung Cancer. In. Chicago, IL: American Lung Association; 2019.
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Background] United States Preventive Services Task Force. Final recommendation statement: Lung cancer screening (updated). https://www.uspreventiveservicestaskforce.org/uspstf/recommendation/lung-cancer-screening. Updated March 9, 2021. Accessed February 21, 2024.
- [Background] Carter-Harris L, Ceppa DP, Hanna N, Rawl SM. Lung cancer screening: what do long-term smokers know and believe? Health Expect. 2017 Feb;20(1):59-68. doi: 10.1111/hex.12433. Epub 2015 Dec 23. PMID 26701339
- [Background] Carter-Harris L, Brandzel S, Wernli KJ, Roth JA, Buist DSM. A qualitative study exploring why individuals opt out of lung cancer screening. Fam Pract. 2017 Apr 1;34(2):239-244. doi: 10.1093/fampra/cmw146. PMID 28122849
- [Background] Carter-Harris L, Slaven JE Jr, Monahan PO, Shedd-Steele R, Hanna N, Rawl SM. Understanding lung cancer screening behavior: Racial, gender, and geographic differences among Indiana long-term smokers. Prev Med Rep. 2018 Feb 3;10:49-54. doi: 10.1016/j.pmedr.2018.01.018. eCollection 2018 Jun. PMID 29552458
- [Background] Carter-Harris L, Slaven JE 2nd, Monahan PO, Draucker CB, Vode E, Rawl SM. Understanding lung cancer screening behaviour using path analysis. J Med Screen. 2020 Jun;27(2):105-112. doi: 10.1177/0969141319876961. Epub 2019 Sep 24. PMID 31550991
- [Background] Draucker CB, Rawl SM, Vode E, Carter-Harris L. Understanding the decision to screen for lung cancer or not: A qualitative analysis. Health Expect. 2019 Dec;22(6):1314-1321. doi: 10.1111/hex.12975. Epub 2019 Sep 27. PMID 31560837
- [Background] De Marchis EH, Brown E, Aceves B, et al. State of the Science of Screening in Healthcare Settings. Social Interventions Research & Evaluation Network, 2022.
- [Background] Albada A, Ausems MG, Bensing JM, van Dulmen S. Tailored information about cancer risk and screening: a systematic review. Patient Educ Couns. 2009 Nov;77(2):155-71. doi: 10.1016/j.pec.2009.03.005. Epub 2009 Apr 18. PMID 19376676
- [Background] Krebs P, Prochaska JO, Rossi JS. A meta-analysis of computer-tailored interventions for health behavior change. Prev Med. 2010 Sep-Oct;51(3-4):214-21. doi: 10.1016/j.ypmed.2010.06.004. Epub 2010 Jun 15. PMID 20558196
- [Background] Kreuter M, Farrell D, Olevitch L, et al. Tailoring health messages: Customizing communication with computer technology. Mahwah, NJ, US: Lawrence Erlbaum Associates Publishers; 2000.
- [Background] Rawl SM, Skinner CS, Perkins SM, Springston J, Wang HL, Russell KM, Tong Y, Gebregziabher N, Krier C, Smith-Howell E, Brady-Watts T, Myers LJ, Ballard D, Rhyant B, Willis DR, Imperiale TF, Champion VL. Computer-delivered tailored intervention improves colon cancer screening knowledge and health beliefs of African-Americans. Health Educ Res. 2012 Oct;27(5):868-85. doi: 10.1093/her/cys094. Epub 2012 Aug 27. PMID 22926008
- [Background] Ruffin MT 4th, Fetters MD, Jimbo M. Preference-based electronic decision aid to promote colorectal cancer screening: results of a randomized controlled trial. Prev Med. 2007 Oct;45(4):267-73. doi: 10.1016/j.ypmed.2007.07.003. Epub 2007 Jul 14. PMID 17689600
- [Background] Ahmad F, Cameron JI, Stewart DE. A tailored intervention to promote breast cancer screening among South Asian immigrant women. Soc Sci Med. 2005 Feb;60(3):575-86. doi: 10.1016/j.socscimed.2004.05.018. PMID 15550305
- [Background] Champion V, Foster JL, Menon U. Tailoring interventions for health behavior change in breast cancer screening. Cancer Pract. 1997 Sep-Oct;5(5):283-8. PMID 9341350
- [Background] Carter-Harris L, Comer RS, Slaven Ii JE, Monahan PO, Vode E, Hanna NH, Ceppa DP, Rawl SM. Computer-Tailored Decision Support Tool for Lung Cancer Screening: Community-Based Pilot Randomized Controlled Trial. J Med Internet Res. 2020 Nov 3;22(11):e17050. doi: 10.2196/17050. PMID 33141096
- [Background] Carter-Harris L, Comer RS, Goyal A, Vode EC, Hanna N, Ceppa D, Rawl SM. Development and Usability Testing of a Computer-Tailored Decision Support Tool for Lung Cancer Screening: Study Protocol. JMIR Res Protoc. 2017 Nov 16;6(11):e225. doi: 10.2196/resprot.8694. PMID 29146565
- [Background] Carter-Harris L, Davis LL, Rawl SM. Lung Cancer Screening Participation: Developing a Conceptual Model to Guide Research. Res Theory Nurs Pract. 2016 Nov 1;30(4):333-352. doi: 10.1891/1541-6577.30.4.333. PMID 28304262
- [Background] Lau YK, Caverly TJ, Cherng ST, Cao P, West M, Arenberg D, Meza R. Development and validation of a personalized, web-based decision aid for lung cancer screening using mixed methods: a study protocol. JMIR Res Protoc. 2014 Dec 19;3(4):e78. doi: 10.2196/resprot.4039. PMID 25532218
- [Background] Memorial Sloan Kettering Cancer Center, Lung cancer screening decision tool. http://nomograms.mskcc.org/Lung/Screening.aspx. Accessed June 20, 2024.
- [Background] Chen Y, Marcus MW, Niaz A, et al My Lung Risk: a user-friendly, web-based calculator for risk assessment of lung cancer based on the validated Liverpool Lung Project risk prediction model. International Journal of Health Promotion and Education. 2014;52(3):144-152.
- [Background] Volk RJ, Linder SK, Leal VB, Rabius V, Cinciripini PM, Kamath GR, Munden RF, Bevers TB. Feasibility of a patient decision aid about lung cancer screening with low-dose computed tomography. Prev Med. 2014 May;62:60-3. doi: 10.1016/j.ypmed.2014.02.006. Epub 2014 Feb 8. PMID 24518006
- [Background] Veterans Health Administration, Screening for lung cancer pamphlet. 2020. http://www.prevention.va.gov/docs/LungCancerScreeningHandout.pdf. Accessed June 20, 2024.
- [Background] Dharod A, Bellinger C, Foley K, Case LD, Miller D. The Reach and Feasibility of an Interactive Lung Cancer Screening Decision Aid Delivered by Patient Portal. Appl Clin Inform. 2019 Jan;10(1):19-27. doi: 10.1055/s-0038-1676807. Epub 2019 Jan 9. PMID 30625501
- [Background] Chew LD, Bradley KA, Boyko EJ. Brief questions to identify patients with inadequate health literacy. Fam Med. 2004 Sep;36(8):588-94. PMID 15343421
- [Background] Thompson HS, Valdimarsdottir HB, Winkel G, Jandorf L, Redd W. The Group-Based Medical Mistrust Scale: psychometric properties and association with breast cancer screening. Prev Med. 2004 Feb;38(2):209-18. doi: 10.1016/j.ypmed.2003.09.041. PMID 14715214
- [Background] Carter-Harris L, Hall LA. Development of a short version of the Cataldo Lung Cancer Stigma Scale. J Psychosoc Oncol. 2014;32(6):665-77. doi: 10.1080/07347332.2014.955238. PMID 25157591
- [Background] Mayo RM, Ureda JR, Parker VG. Importance of fatalism in understanding mammography screening in rural elderly women. J Women Aging. 2001;13(1):57-72. doi: 10.1300/J074v13n01_05. PMID 11217186
- [Background] Carter-Harris L, Slaven JE 2nd, Monohan P, Rawl SM. Development and Psychometric Evaluation of the Lung Cancer Screening Health Belief Scales. Cancer Nurs. 2017 May/Jun;40(3):237-244. doi: 10.1097/NCC.0000000000000386. PMID 27244666
- [Background] Williams DR, Yan Yu, Jackson JS, Anderson NB. Racial Differences in Physical and Mental Health: Socio-economic Status, Stress and Discrimination. J Health Psychol. 1997 Jul;2(3):335-51. doi: 10.1177/135910539700200305. PMID 22013026
- [Background] Weinstein D. The Precaution Adoption Process Model. In: Glanz K, Rimer BK, Viswanath K, eds. Health behavior and health education: Theory, research, and practice, 4th ed. 4th ed. San Francisco, CA, US: Jossey-Bass; 2008:xxxiii-552, pp. 123-147.